CLINICAL TRIAL: NCT06096233
Title: Acute Effect of Exercise on Post-meal Appetite, Appetite-Regulatory Hormones, and Energy Intake in Healthy Men
Brief Title: Effect of Exercise on Appetite in Response to Meals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Northern Border University (Other)
Responsible Party: Principal Investigator, James Dorling, PhD, Lecturer, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200220449
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The participants will not perform any exercise.
- Short Exercise (Experimental): The participants will run on the treadmill for 10 minutes.
  Interventions: Other: Bouts of Exercise
- Prolonged Exercise (Experimental): The participants will run on the treadmill for 30 minutes.
  Interventions: Other: Bouts of Exercise

INTERVENTIONS:
Other: Bouts of Exercise — The participants will run on the treadmill for 10 minutes (short) or 30 minutes (prolonged).
  Arms: Prolonged Exercise; Short Exercise

SUMMARY:
This clinical trial's primary aim is to investigate the acute effect of two exercise bouts (short [10 minutes] and long [30 minutes]) on appetite and appetite-regulatory hormone responses to a standard meal test. The secondary aim is to investigate when the changes in appetite and appetite-regulatory hormones occur during exercise. As an exploratory aim, the researchers will test if the two exercise bouts influence ad libitum energy intake in the periods after the standard meal test. The researchers will compare three groups (control, short exercise, and prolonged exercise) to see if the exercise bouts affect appetite, appetite-regulatory hormones, and energy intake in healthy men.

DETAILED DESCRIPTION:
Study Design

Screening visit Before conducting the main experiments, the participants will attend a screening visit where consent will be obtained, and they will complete questionnaires to assess health, food preferences, and physical activity. The researchers will then measure the participants' height, weight, waist circumference, and body composition.

After the researchers confirm the eligibility criteria, participants will take part in two treadmill tests to establish maximum oxygen uptake test (V̇O2 max) (Broom et al. 2017).

Experimental design After the screening visit, the participants will complete three main experiments (control, short high-intensity exercise, and prolonged high-intensity exercise) in a counter-balanced design. All experiments began at ~0930, following an overnight fast of at least 10 hours. Participants will consume a prescribed meal in the evening before each main experiment. Following this meal, participants are only allowed to drink water until the start of the main experiments.

At the beginning of the exercise conditions, participants will run on the treadmill for 10 minutes (short) or 30 minutes (prolonged) at a speed estimated to elicit a 75% V̇O2 peak, followed by rest in the laboratory. In the control condition, the researchers will follow the same protocols except that the participants will not perform any exercise. The participants will have a standardized meal after exercise and then an ad libitum buffet meal afterward.

During each experiment, the researchers will assess appetite ratings using 100 mm visual analog scales (Flint et al. 2000). The researchers will also collect blood samples to examine ghrelin, peptide YY, glucagon-like peptide 1, and possibly other blood-borne measures.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years or older.
* Have stable body mass for at least six months (within ±2 kg).

Exclusion Criteria:

* Females
* People who are younger than 18 or older than 65 years old.
* Have food allergies.
* Have significant contraindications to exercise (e.g., an injury that would inhibit running).
* Smoking.
* Suffering from metabolic health issues, e.g., history of diabetes, cardiovascular disease, or eating disorders.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Change in Peptide-YY (PYY) | At 0 (baseline), 0.167, 0.5, 1, 1.5, 2, 3, and 4 hours
  Blood samples will be drawn at different time points during the trial to measure the change in PYY blood levels. Area under the plasma concentration versus time curve (AUC) of PYY will be calculated using the trapezoidal rule.
Change in Ghrelin | At 0 (baseline), 0.167, 0.5, 1, 1.5, 2, 3, and 4 hours
  Blood samples will be drawn at different time points during the trial to measure the change in ghrelin blood levels. Area under the plasma concentration versus time curve (AUC) of ghrelin will be calculated using the trapezoidal rule.
Change in Glucagon-Like Peptide-1 (GLP-1) | At 0 (baseline), 0.167, 0.5, 1, 1.5, 2, 3, and 4 hours
  Blood samples will be drawn at different time points during the trial to measure the change in GLP-1 blood levels. Area under the plasma concentration versus time curve (AUC) of GLP-1 will be calculated using the trapezoidal rule.
Change in subjective appetite sensations | At 0 (baseline), 0.167, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 5.5, and 6 hours
  The subjective appetite sensations will be assessed using 100 mm visual analog scales (VAS) to measure appetite sensations (hunger, satiety, fullness, prospective food consumption, and desire to eat). The VAS are 100 mm long, with words anchored at each end expressing the most positive and negative ratings. Scores for each appetite construct range from 0-100.

SECONDARY OUTCOMES:
Energy Intake | At 5 hours
  To determine the amount of each food item consumed, we will measure the difference in weight between before and after the meal. We will use manufacturer details to determine energy consumption.
Macro-nutrient Intake | At 5 hours
  To determine the amount of each food item consumed, we will measure the difference in weight between before and after the meal. We will use manufacturer details to determine macronutrient consumption

CONTACTS AND LOCATIONS:
Overall Officials: James Dorling, PhD, Principal Investigator — University of Glasgow
Locations (1):
- New Lister Building at Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The stored data will be anonymous and follow the guidelines of the General Data Protection Regulation enforced in May 2018. Hard copies of participant information forms, including consent forms and dietary intake records, will be kept in locked filing cabinets. Keys to the filing cabinets will only be available to the primary investigator. All databases will be password protected and stored on a university computer with firewalls.
  Participants' identifiable data will be stored in a locked cabinet. Digital data will be stored anonymously within the server of the University of Glasgow.
  This project's Principal Investigator will be responsible for sharing the research data.
  Data will be preserved in Enlighten, the official online repository of Glasgow University's research output.
Time Frame: The data will be available when the study is completed.
  Data will be preserved for 10 years.
Access Criteria: Data will be shared via the repository deposit (Enlighten). Only signatories of end-user agreements can access and use shared data.

REFERENCES:
- [Background] Broom DR, Miyashita M, Wasse LK, Pulsford R, King JA, Thackray AE, Stensel DJ. Acute effect of exercise intensity and duration on acylated ghrelin and hunger in men. J Endocrinol. 2017 Mar;232(3):411-422. doi: 10.1530/JOE-16-0561. Epub 2016 Dec 20. PMID 27999089
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749